CLINICAL TRIAL: NCT06183931
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Amyloid Depleter ALXN2220 in Adult Participants With Transthyretin Amyloid Cardiomyopathy (ATTR-CM)
Brief Title: Study of ALXN2220 Versus Placebo in Adults With ATTR-CM
Acronym: DepleTTR-CM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6810C00001; ALXN2220-ATTRCM-301 (Other: Alexion)
Record Dates: First submitted 2023-11-15; First posted 2023-12-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Transthyretin Amyloid Cardiomyopathy
Keywords: Amyloid Depleter; ALXN2220; All-cause mortality (ACM); Cardiovascular (CV); Transthyretin Amyloid Cardiomyopathy; Transthyretin amyloid (ATTR); Transthyretin (TTR); N-terminal pro b-type natriuretic peptide (NT-proBNP); NT-proBNP; Amyloidosis; ATTR-CM
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALXN2220 (Experimental): Participants will receive weight-based dose of ALXN2220 via intravenous (IV) infusion every 4 weeks (q4w) for at least 24 months up to a maximum of 48 months.
  Interventions: Drug: ALXN2220
- Placebo (Placebo Comparator): Participants will receive placebo via IV infusion q4w for at least 24 months up to a maximum of 48 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALXN2220 — Participants will receive ALXN2220 via IV infusion.
  Arms: ALXN2220
Drug: Placebo — Participants will receive placebo via IV infusion.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to access the efficacy of ALXN2220 in the treatment of adult participants with ATTR-CM by evaluating the difference between the ALXN2220 and placebo groups as assessed by the total occurrences of all-cause mortality (ACM) and cardiovascular (CV) clinical events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ATTR-CM with either wild-type or variant TTR genotype
* End-diastolic interventricular septal wall thickness ≥ 12 mm on echocardiography measured at Screening
* NT-proBNP > 2000 pg/mL at Screening
* Treatment with a loop diuretic for at least 30 days prior to Screening
* History of heart failure NYHA Class II-IV at Screening
* Life expectancy of ≥ 6 months as per the Investigator's judgment
* Males and females of childbearing ability must use contraception

Exclusion Criteria:

* Known leptomeningeal amyloidosis
* Known light chain (AL) or secondary amyloidosis (AA), or any other form of systemic amyloidosis
* Acute coronary syndrome, unstable angina, stroke, transient ischemic attack, coronary revascularization, cardiac device implantation, cardiac valve repair, or major surgery within 3 months of Screening
* Uncontrolled clinically significant cardiac arrhythmia, per Investigator's assessment
* LVEF < 30% on echocardiography
* Renal failure requiring dialysis or an eGFR < 20 mL/min/1.73 m2 at Screening
* Polyneuropathy with PND score IV

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1181 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2027-06-07 (Estimated); Study Completion 2027-10-05 (Estimated)

PRIMARY OUTCOMES:
Total Occurrence of ACM and CV clinical events during the Blinded Treatment Period | Baseline up to the end study (up to Month 48)

SECONDARY OUTCOMES:
Change From Baseline in Kansas City Cardiomyopathy Questionnaire-Overall Score (KCCQ-OS) at Month 24 | Baseline, Month 24
Time to CV-related Mortality | Baseline up to the end of study (up to Month 48)
Change from Baseline in Six-minute Walk Test (6MWT) at Month 24 | Baseline, Month 24
Total Occurrences of CV Clinical Events | Baseline up to the end of study (up to Month 48)
Time to ACM | Baseline up to the end of study (up to Month 48)

CONTACTS AND LOCATIONS:
Locations (185):
- United States (33):
  - Research Site, Irvine, California
  - Research Site, La Jolla, California
  - Research Site, Palo Alto, California
  - Research Site, San Francisco, California
  - Research Site, Aurora, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Weston, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Boston, Massachusetts
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Stony Brook, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Danville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Falls Church, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
- Australia (7):
  - Research Site, Bedford Park
  - Research Site, Box Hill
  - Research Site, Brisbane
  - Research Site, Darlinghurst
  - Research Site, Joondalup
  - Research Site, Melbourne
  - Research Site, Westmead
- Austria (4):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Vienna
  - Research Site, Wels
- Belgium (3):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Genk
- Brazil (7):
  - Research Site, Aracaju
  - Research Site, Campinas
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Rimouski, Quebec
- China (16):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
- Research Site, Prague, Czechia
- Denmark (2):
  - Research Site, Aarhus
  - Research Site, Odense C
- France (11):
  - Research Site, Bron
  - Research Site, Chambray-lès-Tours
  - Research Site, Créteil
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Poitiers
  - Research Site, Rennes
  - Research Site, Saint-Herblain
  - Research Site, Toulouse
- Germany (13):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Essen
  - Research Site, Giessen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Homburg
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, München
  - Research Site, Münster
  - Research Site, Würzburg
- Research Site, Athens, Greece
- Research Site, Dublin, Ireland
- Israel (5):
  - Research Site, Beer Yaakov
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Rehovot
- Italy (13):
  - Research Site, Bologna
  - Research Site, Ferrara
  - Research Site, Florence
  - Research Site, Forlì
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Torino
  - Research Site, Trieste
- Japan (8):
  - Research Site, Bunkyō City
  - Research Site, Kumamoto
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Matsumoto-shi
  - Research Site, Sapporo
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
- Netherlands (4):
  - Research Site, Groningen
  - Research Site, Maastricht
  - Research Site, Rotterdam
  - Research Site, Utrecht
- Norway (3):
  - Research Site, Lørenskog
  - Research Site, Oslo
  - Research Site, Trondheim
- Poland (3):
  - Research Site, Gdansk
  - Research Site, Poznan
  - Research Site, Warsaw
- South Korea (3):
  - Research Site, Busan
  - Research Site, Seoul
  - Research Site, Wŏnju
- Spain (13):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, El Palmar
  - Research Site, Jaén
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
  - Research Site, Pamplona
  - Research Site, Salamanca
  - Research Site, Santiago de Compostela-Coruña
  - Research Site, Valencia
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Skellefteå
  - Research Site, Stockholm
- Switzerland (5):
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Lucerne
  - Research Site, Sankt Gallen
  - Research Site, Zurich
- Taiwan (3):
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Dinar
  - Research Site, Eskişehir
  - Research Site, Istanbul
  - Research Site, Mersin
- United Kingdom (6):
  - Research Site, Birmingham
  - Research Site, Cardiff
  - Research Site, Glasgow
  - Research Site, Hexham
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR